CLINICAL TRIAL: NCT02503449
Title: Multi-center Clinical Trial of Pulmonary Cryptococcosis in China
Brief Title: Clinical Trial of Pulmonary Cryptococcosis in China
Acronym: MCTOPCIC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhixin Liang (Other)
Collaborators: Chinese PLA General Hospital (Other); Beijing Chao Yang Hospital (Other); Ministry of Health, China (Other Government); Peking University Third Hospital (Other); Tianjin Medical University General Hospital (Other); First Hospital of China Medical University (Other); Shengjing Hospital (Other); Second Hospital of Jilin University (Other); Shandong Provincial Hospital (Other Government); Huadong Hospital (Other); Nanjing PLA General Hospital (Other); Fuzhou General Hospital (Other); Guangzhou Institute of Respiratory Disease (Other); Wuhan TongJi Hospital (Other); Xi'an Jiaotong University (Other); Guizhou Provincial People's Hospital (Other); Shenyang Military General Hospital (Unknown); The Second Hospital of Hebei Medical University (Other); Xiangya Hospital of Central South University (Other); Fujian Provincial Hospital (Other); Fuzhou Pulmonary Hospital of Fujian (Other); Southwest Hospital, China (Other); First Affiliated Hospital of Zhejiang University (Other); Wenzhou Medical University (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Longyan City First Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhixin Liang, Chinese Medical Association of respiratory diseases, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: LYN-316
Record Dates: First submitted 2014-12-28; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Cryptococcosis
Keywords: Pulmonary Cryptococcosis
MeSH Terms: conditions — Cryptococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — sputum,whole blood,pleural effusion,lung tissue,cerebrospinal fluid,fungus(smear examination,culture and identification,antigen detection,drug sensitive test)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study:1.Improve the understanding of the risk factors of pulmonary cryptococcosis;2.Improve the awareness of pulmonary cryptococcosis clinical and imaging manifestations;3.Grasp pulmonary cryptococcosis patients of clinical and imaging manifestations in different conditions;4.Learn about antibacterial activity of antifungal drugs for cryptococcosis in China.

DETAILED DESCRIPTION:
1. Patients corresponding to inclusion criteria and obtaining informed consent are included in the research in department of respiration ward in cooperative hospitals.
2. Relevant case report forms are created in this study.
3. Basic information such as age,weight and height is recorded in selected cases.Clinical manifestations,risk factors,laboratory examination,imaging examination,etiological examination and histopathological examination are also recorded in selected cases by case report forms.In addition,antifungal treatment is recorded including name,dose,time of starting treatment and terminate treatment.Causes of terminate treatment and curative effect evaluation should be analysed.
4. Statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients possess clinical or imaging manifestations of pulmonary infections,with any of the results(by one of following conditions) by microbiological examination or histopathologic examination

1. Cryptococcal capsular polysaccharide antigen of blood or pleural effusion is positive
2. Cryptococcus（fungus culture) is discovered by lower respiratory tract specimens
3. Cryptococcus（pleural effusions culture) is discovered by pleural effusions collected under sterile condition
4. Cryptococcus（pus culture) is discovered by pus smear out of pulmonary infections in disseminated infection patients
5. Cryptococcus（blood culture) is discovered by microscopy of specimens of blood smear
6. Cryptococcus is discovered by culturing of the pathological tissue specimens in aseptic condition
7. Cryptococcal capsular budding yeast with inflammatory reaction is discovered by histopathological examination,cell pathology examination or microscopic examination in aseptic condition

Exclusion Criteria:

1. Patients suffer from acquired immune deficiency syndrome
2. Patients or their legal guardians request to withdraw the clinical research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Improve the understanding of the risk factors of pulmonary cryptococcosis.
  2. Improve the awareness of pulmonary cryptococcosis clinical and imaging manifestations.
  3. Grasp pulmonary cryptococcosis patients of clinical and imaging manifestations in different conditions.
  4. Learn about antibacterial activity of antifungal drugs for cryptococcosis in China.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
differences in clinical manifestations of pulmonary cryptococcosis | 30 days
  Methods including laboratory examination(routine blood test),imaging examination(chest CT),scoring system(APACHE II score)

SECONDARY OUTCOMES:
treatment of pulmonary cryptococcosis | 30 days
  Efficacy as measured by recording dose and time of therapy for antifungal agents

CONTACTS AND LOCATIONS:
Overall Officials: Zhixin Liang, Doctor, Study Director — Chinese PLA General Hospital; Zhen Wang, Principal Investigator — Beijing Chao Yang Hospital; Yanming Li, Principal Investigator — Ministry of Health, China; Lina Sun, Principal Investigator — Peking University Third Hospital; Jie Cao, Principal Investigator — Tianjin Medical University General Hospital; Yunzhuo Chu, Principal Investigator — First Hospital of China Medical University; Zhijie Zhang, Principal Investigator — Shengjing Hospital; Yufen Jin, Principal Investigator — Second Hospital of Jilin University; Xiaobin Ma, Principal Investigator — Shandong Provincial Hospital; Yanping Zhu, Principal Investigator — Huadong Hospital; Xin Su, Principal Investigator — Nanjing PLA General Hospital; Guoxiang Lai, Principal Investigator — Fuzhou General Hospital; Feng Ye, Principal Investigator — Guangzhou Institute of Respiratory Disease; Shengdao Xiong, Principal Investigator — Wuhan TongJi Hospital; Lan Yang, Principal Investigator — Xi'an Jiaotong University; Hong Yu, Principal Investigator — Guizhou Provincial People's Hospital; wencheng Xue, Principal Investigator — Shenyang Military General Hospital; Yadong Yuan, Principal Investigator — The Second Hospital of Hebei Medical University; Chengping Hu, Principal Investigator — Xiangya Hospital of Central South University; Baosong Xie, Principal Investigator — Fujian Provincial Hospital; Xiaohong Chen, Principal Investigator — Fuzhou Pulmonary Hospital of Fujian; Xiangdong Zhou, Principal Investigator — Southwest Hospital, China; Wenjiang Ma, Principal Investigator — First Affiliated Hospital of Zhejiang University; Yuping Li, Principal Investigator — Wenzhou Medical University; Hongni Jiang, Principal Investigator — Shanghai Zhongshan Hospital; Wei Bai, Principal Investigator — The First Affiliated Hospital of Nanchang University; Sucheng Zhong, Principal Investigator — Longyan City First Hospital